CLINICAL TRIAL: NCT07136493
Title: Evaluation of Circulating Tumor DNA Based Minimal Residual Disease Detection in Early Stage Breast Cancer Patients: A Prospective Study
Brief Title: Circulating Tumor DNA Based Minimal Residual Disease Detection for Patients With Early-Stage Breast Cancer
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 24463; NCI-2025-05431 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24463 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-08-10; First posted 2025-08-22 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Estrogen Receptor-Positive Breast Carcinoma; HER2-Negative Breast Carcinoma; HER2-Positive Breast Carcinoma; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (blood collection for ctDNA testing - 1) (Experimental): Patients undergo collection of blood samples for ctDNA testing at 14-21 days post cycle 1, day 1 of SOC neoadjuvant chemotherapy, on the day of SOC surgery, at 3-6 weeks after SOC surgery, at 1-2 weeks after SOC adjuvant radiation therapy (if receiving), at 2-4 weeks after SOC adjuvant systemic therapy (if receiving), every 3 months for 1 year after surgery, and then every 6 months up to year 3 after surgery. Patients may also undergo collection of tumor tissue during SOC surgery on study.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review; Other: Survey Administration
- Cohort 2 (blood collection for ctDNA testing -2) (Experimental): Patients undergo collection of blood samples for ctDNA testing on the day of SOC surgery, at 3-6 weeks after SOC surgery, at 1-2 weeks after SOC adjuvant radiation therapy (if receiving), at 2-4 weeks after SOC adjuvant systemic therapy (if receiving), every 3 months for 1 year after surgery, and then every 6 months up to year 3 after surgery. Patients may also undergo collection of tumor tissue during SOC surgery on study.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review; Other: Survey Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples for ctDNA testing
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Biospecimen Collection — Undergo possible collection of tissue
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Electronic Health Record Review — Ancillary studies
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial studies how well circulating tumor deoxyribonucleic acid (ctDNA) based minimal residual disease (MRD) detection works for patients with early-stage breast cancer. MRD refers to a very small number of tumor cells that remain in the body during or after treatment. ctDNA refers to small pieces of DNA that are released into a person's blood by tumor cells as they die. Management of patients after cancer surgery remains a clinical dilemma, particularly for cancer detected at earlier stages as many patients are cured by surgery alone. This results in very large clinical trials required to demonstrate a modest benefit from treatment. Using ctDNA MRD testing in early-stage breast cancer patients receiving standard treatment may help researchers identify groups that would benefit from additional therapy, leading to better outcomes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the pathologic response rate and presence of ctDNA post-neoadjuvant therapy in stage I-III breast cancer patients receiving neoadjuvant systemic therapy followed by curative-intent surgical resection, separately for Subgroup 1A: human epidermal growth factor receptor 2 positive (HER2+) (any estrogen receptor [ER]/progesterone receptor [PR] status) and Subgroup 1B: triple negative breast cancer (TNBC). (Cohort 1) II. To determine ctDNA detectability before and after curative-intent surgical resection in Cohort 2 ER+/any progesterone receptor (PR)/HER2- stage I-III breast cancer patients. (Cohort 2)

SECONDARY OBJECTIVES:

I. To determine ctDNA detectability before and after adjuvant chemotherapy and/or radiation therapy, by cohort and subgroup.

II. To determine ctDNA detectability during the follow-up period of up to 3 years after definitive treatment, by cohort and subgroup.

III. To describe, by cohort and subgroup, the association between detectable ctDNA measured post-neoadjuvant treatment and post-surgery with recurrence free survival (RFS).

IV. To describe, by cohort and subgroup, ctDNA levels at baseline and during neoadjuvant treatment and their association with clinical and pathologic response.

V. To describe, by cohort and subgroup, changes in ctDNA levels during systemic treatment (neoadjuvant and adjuvant) and association with clinical response determined radiographically.

VI. To describe, by cohort and subgroup, the difference in time between ctDNA detection (molecular recurrence) and radiographic evidence of disease recurrence following definitive treatment among patients who achieved undetectable ctDNA levels after surgery.

EXPLORATORY OBJECTIVE:

I. To explore the performance of up to two cancer detection assays - BestSEEK and enACT - in development by Dr. Tomasetti at TGen and City of Hope.

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT 1: Patients undergo collection of blood samples for ctDNA testing at 14-21 days post cycle 1, day 1 of standard of care (SOC) neoadjuvant chemotherapy, on the day of SOC surgery, at 3-6 weeks after SOC surgery, at 1-2 weeks after SOC adjuvant radiation therapy (if receiving), at 2-4 weeks after SOC adjuvant systemic therapy (if receiving), every 3 months for 1 year after surgery, and then every 6 months up to year 3 after surgery. Patients may also undergo collection of tumor tissue during SOC surgery on study.

COHORT 2: Patients undergo collection of blood samples for ctDNA testing on the day of SOC surgery, at 3-6 weeks after SOC surgery, at 1-2 weeks after SOC adjuvant radiation therapy (if receiving), at 2-4 weeks after SOC adjuvant systemic therapy (if receiving), every 3 months for 1 year after surgery, and then every 6 months up to year 3 after surgery. Patients may also undergo collection of tumor tissue during SOC surgery on study.

ELIGIBILITY:
Inclusion Criteria:

* Documented written informed consent of the participant
* Age ≥ 18 years
* Diagnosis of stage I-III breast cancer (any gender)
* Malignancy must be epithelial. Non-epithelial breast malignancies such as lymphoma or sarcoma are not allowed
* Willingness to:

  * Provide blood samples
  * Provide archival tumor tissue sample (only necessary for Cohort 2 if analysis of surgical tissue was not successful)
  * Provide tumor tissue sample from resection/surgery (only necessary for Cohort 1 if analysis of surgical tissue was not successful)
  * Permit medical record review
* Fall into one of the following categories defined below: Cohort 1, Subgroup A or B OR Cohort 2
* COHORT 1: Must have archival diagnostic tissue available
* COHORT 1: Scheduled to undergo, but has not yet begun, neoadjuvant systemic therapy followed by curative resection
* COHORT 1 (Subgroup A): HER2+ by current American Society of Clinical Oncology (ASCO)/College of American Pathologist (CAP) guidelines (any ER/PR status)
* COHORT 1 (Subgroup B): Triple negative (ER, PR and HER2 negative). Defined as ER and PR ≤ 10% by immunohistochemistry (IHC) and HER2 negative, by current ASCO/CAP guidelines
* COHORT 2: Scheduled to undergo upfront curative surgical resection with or without adjuvant chemotherapy followed by adjuvant endocrine therapy
* COHORT 2: ER+/any PR/HER2- (ER positive defined as ER > 10% by IHC)

Exclusion Criteria:

* Ductal carcinoma in situ
* Inability to safely provide sequential blood samples
* Prior or concurrent invasive malignancy (unless disease free > 5 years)
* An employee who is under the direct/ indirect supervision of the principal investigator (PI)/ a co-investigator/ the study manager
* A direct study team member
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients that achieve a pathologic complete response and are circulating tumor deoxyribonucleic acid (ctDNA) detectable (Cohort 1) | Up to 3 years after standard of care (SOC) surgery
  Baseline characteristics will be compared using the K-sample equality-of-medians test with continuity correction and the two-sample test of proportions. Cox proportional-hazards models, with the exact partial likelihood method to handle tied event times and adjusting for post-baseline ctDNA (negative versus positive), baseline tumor marker (not elevated versus elevated), and tumor stage as pre-specified confounders. Other confounders will be adjusted for as appropriate.
ctDNA detection rate (Cohort 2) | Before and after SOC surgery (up to 3 years)
  Baseline characteristics will be compared using the K-sample equality-of-medians test with continuity correction and the two-sample test of proportions. Cox proportional-hazards models, with the exact partial likelihood method to handle tied event times and adjusting for post-baseline ctDNA (negative versus positive), baseline tumor marker (not elevated versus elevated), and tumor stage as pre-specified confounders. Other confounders will be adjusted for as appropriate.

SECONDARY OUTCOMES:
ctDNA detection rate 1 | Before and after adjuvant chemotherapy and/or radiation therapy (up to 3 years)
  Baseline characteristics will be compared using the K-sample equality-of-medians test with continuity correction and the two-sample test of proportions. Cox proportional-hazards models, with the exact partial likelihood method to handle tied event times and adjusting for post-baseline ctDNA (negative versus positive), baseline tumor marker (not elevated versus elevated), and tumor stage as pre-specified confounders. Other confounders will be adjusted for as appropriate.
ctDNA detection rate 2 | Up to 3 years post-definitive treatment
  Baseline characteristics will be compared using the K-sample equality-of-medians test with continuity correction and the two-sample test of proportions. Cox proportional-hazards models, with the exact partial likelihood method to handle tied event times and adjusting for post-baseline ctDNA (negative versus positive), baseline tumor marker (not elevated versus elevated), and tumor stage as pre-specified confounders. Other confounders will be adjusted for as appropriate.
Recurrence free survival (RFS) | Post-neoadjuvant treatment and post-surgery (up to 3 years)
  Baseline characteristics will be compared using the K-sample equality-of-medians test with continuity correction and the two-sample test of proportions. RFS will be compared using univariate and multivariate Cox proportional-hazards models, with the exact partial likelihood method to handle tied event times and adjusting for post-baseline ctDNA (negative versus positive), baseline tumor marker (not elevated versus elevated), and tumor stage as pre-specified confounders.
ctDNA level | Up to 3 years after SOC surgery
  Baseline characteristics will be compared using the K-sample equality-of-medians test with continuity correction and the two-sample test of proportions. Cox proportional-hazards models, with the exact partial likelihood method to handle tied event times and adjusting for post-baseline ctDNA (negative versus positive), baseline tumor marker (not elevated versus elevated), and tumor stage as pre-specified confounders. Other confounders will be adjusted for as appropriate.
Rate of concordance between ctDNA changes on systemic treatment and clinical response | Up to 3 years after SOC surgery
  Agreement in change in ctDNA and radiologic response will be assessed based on increase/decrease/clearance in ctDNA and response of complete response/partial response/stable disease or progressive disease. Data visualization may be used to help understand changes in ctDNA over time by patient, cohort, subgroup, and treatment type (e.g., a spider plot).
Difference in time between ctDNA detection date and radiographic disease progression date | Up to 3 years after SOC surgery
  In patients with undetectable ctDNA levels directly following surgery, the time when ctDNA is first detected during follow-up will be identified and the proximity of this time to radiographic evidence of disease will be calculated. Kaplan-Meier will be used to estimate the median time interval for detection of disease, as we anticipate censoring to occur with this endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Jose G Bazan, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (5):
- United States (5):
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope at Irvine Lennar, Irvine, California
  - City of Hope Atlanta Cancer Center, Newnan, Georgia
  - City of Hope at Chicago, Zion, Illinois